CLINICAL TRIAL: NCT01695785
Title: Perception of Physical Exertion in Healthy Weight and Obese Adolescents: A Pilot Study
Brief Title: Perception of Physical Exertion in Healthy Weight and Obese Adolescents
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Connie Tompkins, PhD, Assistant Professor, University of Vermont
Other Study IDs: M12-079
Record Dates: First submitted 2012-09-24; First posted 2012-09-28 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Physiological Response to Exercise; Perception of Exercise Difficulty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy weight: greater than or equal to the 5th to less than the 85th BMI percentile
- Obese: greater than or equal to the 95th BMI percentile

SUMMARY:
Little is known regarding the relationship between perceived and physiological exertion in adolescents. The purpose of this study is to investigate the association between physiological and perceptual markers of effort during exercise and the relationship of these markers to other health-related behaviors in healthy weight and obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy weight (>5th-85th BMI percentile) or obese (>95th BMI percentile)
* male and female adolescents, 13-18 years
* Approval to participate in a submaximal and maximal treadmill test received from the adolescent's pediatrician.

Exclusion Criteria:

* Underweight (<5th BMI percentile)
* overweight (85 - <95th BMI percentile)
* evidence/reporting of significant cardiovascular disease, cardiac arrhythmias, liver disease, or the chronic use of medications including diuretics, steroids and adrenergic-stimulating agents.
* Adolescents with emotional problems such as clinical depression or other diagnosed psychological condition and currently use prescription medication for psychological conditions.
* Approval to participate in a submaximal and maximal treadmill test from the adolescent's pediatrician not obtained

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy weight and obese adolescents from the community
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Physiological responses to submaximal and maximal treadmill exercise | 7-10 days
  Physiological responses to submaximal and maximal treadmill exercise will be assessed during the exercise test and immediately upon completion of the exercise test. The submaximal treadmill exercise will take place at visit 1 and the maximal treadmill exercise test will take place at the 2nd and final visit which will occur 7-10 days from the 1st visit. There is no intervention between visits.

SECONDARY OUTCOMES:
Perceptual responses to submaximal and maximal treadmill exercise | 7-10 days
  Perceptual responses to submaximal and maximal treadmill exercise will be assessed during the exercise test and immediately upon completion of the exercise test. The submaximal treadmill exercise will take place at visit 1 and the maximal treadmill exercise test will take place at the 2nd and final visit which will occur 7-10 days from the 1st visit. There is no intervention between visits.

OTHER OUTCOMES:
Physical activity intention | 7 days
  Subjects will be asked how much physical activity they plan or intend to participate in for the next 7 days.
Physical activity behavior | 7 days
  Subjects will be asked how much physical activity they participated in for the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Tompkins, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States